CLINICAL TRIAL: NCT02136784
Title: Analgesic Response to Opioid Analgesics in Buprenorphine-Maintained Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: Indivior Inc. (Industry)
Responsible Party: Principal Investigator, Walter Ling, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 13-001175
Record Dates: First submitted 2014-03-18; First posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Analgesic Response
Keywords: pain; cold presser test; buprenorphine; opioids
MeSH Terms: conditions — Pain | interventions — Morphine; Hydrocodone; Oxycodone; Buprenorphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (7):
- morphine sulfate (Experimental): 30mg, single dose,
  Interventions: Drug: oral tablet placebo
- hydrocodone (Experimental): 10mg single dose
  Interventions: Drug: oral tablet placebo
- hydromorphone HCI (Experimental): 4mg single dose
  Interventions: Drug: oral tablet placebo
- oxycodone (Experimental): 10 mg single dose
  Interventions: Drug: oral tablet placebo
- buprenorphine (Experimental): 4 mg single dose
  Interventions: Drug: sublingual tablet placebo
- oral tablet placebo (Placebo Comparator): single dose
  Interventions: Drug: morphine sulfate; Drug: hydrocodone; Drug: hydromorphone HCI; Drug: oxycodone
- sublingual tablet placebo (Placebo Comparator): single dose
  Interventions: Drug: buprenorphine

INTERVENTIONS:
Drug: morphine sulfate — Participants will receive randomly assigned order of study drug (opioid) and then have 7 days of testing with test days at least 3 days apart. Pain testing will utilize cold pressor test, in which the participant submerges his arm and hand in a bath of ice cold water to determine pain threshold and tolerance.
  Other Names: 30 mg, single dose
  Arms: oral tablet placebo
Drug: hydrocodone — Participants will receive randomly assigned order of study drug (opioid) and then have 7 days of testing with test days at least 3 days apart. Pain testing will utilize cold pressor test, in which the participant submerges his arm and hand in a bath of ice cold water to determine pain threshold and tolerance.
  Other Names: 10mg single dose
  Arms: oral tablet placebo
Drug: hydromorphone HCI — Participants will receive randomly assigned order of study drug (opioid) and then have 7 days of testing with test days at least 3 days apart. Pain testing will utilize cold pressor test, in which the participant submerges his arm and hand in a bath of ice cold water to determine pain threshold and tolerance.
  Other Names: 4 mg single dose
  Arms: oral tablet placebo
Drug: oxycodone — Participants will receive randomly assigned order of study drug (opioid) and then have 7 days of testing with test days at least 3 days apart. Pain testing will utilize cold pressor test, in which the participant submerges his arm and hand in a bath of ice cold water to determine pain threshold and tolerance.
  Other Names: 10 mg single dose
  Arms: oral tablet placebo
Drug: buprenorphine — Participants will receive randomly assigned order of study drug (opioid) and then have 7 days of testing with test days at least 3 days apart. Pain testing will utilize cold pressor test, in which the participant submerges his arm and hand in a bath of ice cold water to determine pain threshold and tolerance.
  Other Names: 4 mg single dose
  Arms: sublingual tablet placebo
Drug: oral tablet placebo — Participants will receive randomly assigned order of study drug (opioid) and then have 7 days of testing with test days at least 3 days apart. Pain testing will utilize cold pressor test, in which the participant submerges his arm and hand in a bath of ice cold water to determine pain threshold and tolerance.
  Other Names: single dose
  Arms: hydrocodone; hydromorphone HCI; morphine sulfate; oxycodone
Drug: sublingual tablet placebo — Participants will receive randomly assigned order of study drug (opioid) and then have 7 days of testing with test days at least 3 days apart. Pain testing will utilize cold pressor test, in which the participant submerges his arm and hand in a bath of ice cold water to determine pain threshold and tolerance.
  Other Names: single dose
  Arms: buprenorphine

SUMMARY:
The aim of this study is to examine the effects of opioid analgesics on acute pain in participants maintained on buprenorphine+naloxone (Suboxone) for opioid use disorders. Seven medication conditions will be tested in a cold pressor test (CPT) paradigm.

DETAILED DESCRIPTION:
Study design is a single-blind examination of the analgesic effects of a single dose of seven test medications provided in an experimental pain paradigm using a cold pressor test (CPT). Test medication conditions include buprenorphine, morphine, hydromorphone, hydrocodone, oxycodone, and two placebo conditions to match test medication formulations (oral tablet, sublingual tablet). Each medication condition will be tested on separate days (seven total days, completing within 12 weeks), with random assignment to order of study medications. After screening, eligible participants will be scheduled for 7 days of testing with test days at least 3 days apart to provide a sufficient medication wash-out period. Pain testing will utilize cold pressor tests (CPT), in which the participant submerges his arm and hand in a bath of ice cold water to determine pain threshold and tolerance. Participants will be given a practice trial to provide familiarity with the test and reduce test anxiety. Two CPTs will occur on each test day, and pre- and post-CPT assessments will be administered. Blood samples will be taken on each test day to measure blood levels of buprenorphine. Daily procedures include: (1) A baseline CPT (BL-CPT), (2) Administration of the test medication (active drug or placebo), (3) CPT administered at the time of maximum drug effect (Tmax-CPT) specific to medication (range 30-120 minutes), (4) Pupillometry conducted at baseline (before BL-CPT), and at time of maximum drug effect (before Tmax-CPT). Each participant will be discharged after clinical determination of the participant's safety and well-being. Testing will continue until twelve trials of each medication condition are completed.

ELIGIBILITY:
Inclusion Criteria:

1. Male, in good general health
2. 20-50 years old
3. Fluent in English
4. Maintained on buprenorphine for at least 3 months
5. Able to complete testing/assessments for 7 test days within 12 weeks
6. Approved for participation by buprenorphine-prescribing physician

Exclusion Criteria:

1. Known hypersensitivity to any of the test opioids
2. Urine test positive for opioids (other than buprenorphine) or other illicit substances
3. Current use of any additional opioid or analgesic medication (other than buprenorphine), medical marijuana, MAOI, tricyclic antidepressant, duloxetine, gabapentin, pregabalin, or other medication considered unsafe or having potential to influence pain perception as determined by study physician.
4. Presence of acute pain condition or planned surgery during the study period
5. Unstable vital signs as determined by the study physician.
6. Current pattern of alcohol, benzodiazepine, or other sedative hypnotic use, as determined by the study medical clinician, which would preclude safe participation in the study;
7. Pending legal action or other situation that might prevent remaining in the area for the duration of the study
8. Current medical or psychiatric condition that could detract from study objectives, place the participant at risk, or interfere with treatment goals

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Pain detection | 7 testing sessions over 12 weeks
  Pain detection is defined as the number of seconds it takes for the participant to feel pain.
Pain tolerance | 7 testing sessions over 12 weeks
  Pain tolerance is defined as the number of seconds it takes before the participant removes his hand from the ice water.

SECONDARY OUTCOMES:
Pupillometry results | 7 testing sessions over 12 weeks
  Examine pupillometry results in the context of administered opioid medications and associated cold pressor tests.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Integrated Substance Abuse Programs Outpatient Clinical Research Center, Los Angeles, California, United States